CLINICAL TRIAL: NCT04461470
Title: 6-Month Outcomes of Pulsed Electro Resonance to Nucleotide Sources Revealing Cell Sensory Experience in Pain Relief, Stress Relief and Anti-ageing Homeostatic Restoration
Brief Title: 6-Month Outcomes of PEMF to Nucleotide Sources Revealing Cell Sensory Experience in Pain Relief, Stress Relief and Anti Ageing Restoration
Acronym: PEMF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: hz Clinic (Industry)
Collaborators: East London Electric Company (Unknown); PropDesk (Unknown); MedCity (Unknown); UCL Partners (Unknown); Imperial College London Partners (Unknown); Health Innovation Network (Unknown)
Responsible Party: Sponsor
Other Study IDs: 7012
Record Dates: First submitted 2020-07-03; First posted 2020-07-08 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-02

CONDITIONS: Pain; Stress; Ageing Signs; Immunity Compromise
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- London: pulsed electro resonance hz 4, hz 3, hz 2, hz 3.5 and residual hz 5
  Interventions: Genetic: epigenetic longitudinal waves
- All United Kingdom: pulsed electro resonance hz 4, hz 3, hz 2, hz 3.5 and residual hz 5
  Interventions: Genetic: epigenetic longitudinal waves

INTERVENTIONS:
Genetic: epigenetic longitudinal waves — force - inducing energies using electromagnetic field(s)
  Other Names: hz

SUMMARY:
Background:

The hz Clinic registry is a programme made of five scheduled cohorts designed to include participants dealing with Immunity compromise, Pain, Ageing and Stress (general and pandemic anxieties) who are to be followed for 6 month to five years in their structured routine of pulsed electro resonance (PEMF) to determine their clinical outcome in the real world, contributing evidence for benchmarking fellow cohort participant variance.

Here we report baseline characteristics, PEMF transfer events and outcomes in participants in the UK. This study serves as a calibration proforma for downstream real world evidence observations of PEMF in the field.

DETAILED DESCRIPTION:
Introduction:

Electro resonance (PEMF) therapy is relatively new, despite the fact that it is considered a gold standard approach in healthcare application.

The base premise of PEMF is to apply field (inducing force) energies to a host, producing a spectrum of physiological benefits (Bagnato et al., 2015). The advantages of PEMF approaches are the vast modalities available in which an inducing force is applied and is configured (low to high hz intensity, frequency and polarity). The disadvantages are, however, dissonances in paradigm trajectory and PEMF seldom interrogation of the in-situ / in-vivo metrics of change in recipient (Funk et al., 2008; Peterchev et al., 2012).

PEMF data in healthcare enables an exercise of compelled judgement(s) across all critical level (pre-clinical, phase I, phase II, phase III, phase IV) system activity. Today there is an apparent disjoint of insight between systems-derived data (imaging) and treatment applied data (remedial action). Some example settings of this include i) electro resonance / surgery as an evidence based tool in clinical decision making (Phelps et al., 2018 and Strauch et al., 2009); ii) in-vitro electro resonance in skin equivalence model (Mitchell et al., 2015 and Mitchell et al., 2016) and bone stimulus model (Ferroni et al., 2018) modelling in-vivo benefit; iii) phase IV anticoagulation and prothrombin ratio 'observations and stratification' using principle component positions, and observing all contributing variances in play (Sawhney et al., 2018).

The unprecedented contribution of pandemic variance (Huang et al., 2020), is heightening a public awareness of how manifold real world evidence is in resolving the insight disjoints. Biomedical problems occur in forms where remote or aseptic application and self observation is paramount to care; particularly in the cases of infection, healing wounds and hydro-electrolyte restoration(s).

In plentiful coverage, PEMF homeostatic benefits on Immunity compromise, Pain, Stress and Ageing are extensively reviewed with Mun et al., (2018); and although the mechanisms of actions are underpinned; our literature search shows that there are seldom real world initiatives, recording wide-spread physiological improvements that PEMF therapy enacts.

Aim:

Here we describe the calibration proforma of PEMF correspondence scoring in longitudinal, physiological and observational outcomes. This study will serve as method development for downstream real world evidence observations of PEMF in the field.

Method:

Ethics statement

All participants provided written informed consent in the online basket checkout at hzclinic.co.uk opting to be therapy subjects. The registry is being conducted in accordance with local regulatory requirements, and the International Conference on Harmonisation-Good Pharmacoepidemiological and Clinical Practice Guidelines.

Procedures and outcomes measures

Baseline data collected at screening included participant characteristics (like age), type of clinical-problem (Stress, Pain, Immunity compromise), date and method of diagnosis if any formal, symptoms, and PEMF treatment (delocalised resonance over nucleotide source inducing post transcription modification (PTM) to ubiquitous properties (U.P.)) 2 hz PTM; 3 hz PTM; 4 hz PTM; 5 hz PTM [request appendix for additional I.P. support].

Data on all components of (and) the McGill Life (Sensory, Affectory, Evaluative, Miscellaneous) Index Chart (recordings) were collected to assess the sensitivities of Pain, Stress, Ageing and Immunity compromise states retrospectively.

hz data were collected using a proprietary electronic case report form (eCRF) captured by trained personnel. Oversight of the operations and data management are managed by the coordinating centre hz Clinic, with supporting entities PropDesk (London, UK) and East London Electric Company (ELEC) (London, UK); and resourcing centres MedCity in conjunction with UCL Partners, Imperial College Health Partners and the Health Innovation Network.

The hz protocol requires that 20% of all eCRFs are monitored against source documentation, that there is an electronic audit trail for all data modifications, and that critical variables are subjected to additional audit (Cohen et al., 2015).

Statistical analysis

This article describes the baseline characteristics, treatment patterns and 6 month outcomes based on national data and for participants included in the UK; data for these analyses were extracted from the registry database on 12th February 2020. Continuous variables are expressed as mean ± standard deviation (SD) and categorical variables as frequency and percentage. Utility of PEMF at baseline was analysed by McGill Life Chart Index scores, calculated retrospectively from the data collected. Participants with missing values were not removed from the study. National normalised ratio (NNR) readings during the 6 months follow up were included in the analysis. We adapted the international normalised ratio (Bonar and Favaloro., 2016) with the acquisition and processing of urine samples for participant metabolome mass fingerprinting and hydration readings as an index, performed (request appendix for additional NNR guidelines). Implausible NNR value of less than 0.8 or greater than 20 were excluded. The distribution of NNR values are described by counts and percentages below, within, and above the therapeutic range, and by the mean, SD, median, and interquartile range (IQR).

Occurrence of major clinical response (primarily, Pain-relief, Stress-relief, anti-oxidation (/ageing) and quenched inflammation) is described using the number of events, the proportion of participants with the event divided by the population at burden at the beginning of the follow-up-period, person-time event rate (per 100 person-years), and 95% confidence interval (CI). We estimated person-year rates using a Poisson model, with the number of events. Only the first occurrences of each event were taken into account. Data analysis was performed at the PropDesk with MatLab (MathsWorks, Massachusetts, USA).

ELIGIBILITY:
Inclusion Criteria:

* Adept to social media / technology uses and convenience of care / health benchmarking

Exclusion Criteria:

* History of cardiovascular issue

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Distinct community regions - United Kingdom, London.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-08-29 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2024-09-12 (Estimated)

PRIMARY OUTCOMES:
Pain alleviation | Imminence - one day
  McGill Index Score 0 - 5
Stress alleviation | Imminence - one day
  McGill Index Score 0 - 5
Anti ageing | Imminence - one day
  McGill Index Score 0 - 5
Inflammation quenching | Imminence - one day
  McGill Index Score 0 - 5

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Davies, Study Chair — East London Electric Company
Locations (1):
- hz Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
researchers can contribute to the cohort and bridge their access to participant-centred data

REFERENCES:
- [Background] Bagnato GL, Miceli G, Marino N, Sciortino D, Bagnato GF. Pulsed electromagnetic fields in knee osteoarthritis: a double blind, placebo-controlled, randomized clinical trial. Rheumatology (Oxford). 2016 Apr;55(4):755-62. doi: 10.1093/rheumatology/kev426. Epub 2015 Dec 24. PMID 26705327
- [Background] Booth CM, Tannock IF. Randomised controlled trials and population-based observational research: partners in the evolution of medical evidence. Br J Cancer. 2014 Feb 4;110(3):551-5. doi: 10.1038/bjc.2013.725. Epub 2014 Jan 14. No abstract available. PMID 24495873
- [Background] Ferroni L, Gardin C, Dolkart O, Salai M, Barak S, Piattelli A, Amir-Barak H, Zavan B. Pulsed electromagnetic fields increase osteogenetic commitment of MSCs via the mTOR pathway in TNF-alpha mediated inflammatory conditions: an in-vitro study. Sci Rep. 2018 Mar 23;8(1):5108. doi: 10.1038/s41598-018-23499-9. PMID 29572540
- [Background] Funk RH. Coupling of pulsed electromagnetic fields (PEMF) therapy to molecular grounds of the cell. Am J Transl Res. 2018 May 15;10(5):1260-1272. eCollection 2018. PMID 29887943
- [Background] Kolifarhood G, Aghaali M, Mozafar Saadati H, Taherpour N, Rahimi S, Izadi N, Hashemi Nazari SS. Epidemiological and Clinical Aspects of COVID-19; a Narrative Review. Arch Acad Emerg Med. 2020 Apr 1;8(1):e41. eCollection 2020. PMID 32259130
- [Background] Mitchell CA, Long H, Donaldson M, Francese S, Clench MR. Lipid changes within the epidermis of living skin equivalents observed across a time-course by MALDI-MS imaging and profiling. Lipids Health Dis. 2015 Aug 5;14:84. doi: 10.1186/s12944-015-0089-z. PMID 26243140
- [Background] Mitchell CA, Donaldson M, Francese S, Clench MR. MALDI MSI analysis of lipid changes in living skin equivalents in response to emollient creams containing palmitoylethanolamide. Methods. 2016 Jul 15;104:93-100. doi: 10.1016/j.ymeth.2016.02.001. Epub 2016 Feb 2. PMID 26845462
- [Background] Mun EJ, Babiker HM, Weinberg U, Kirson ED, Von Hoff DD. Tumor-Treating Fields: A Fourth Modality in Cancer Treatment. Clin Cancer Res. 2018 Jan 15;24(2):266-275. doi: 10.1158/1078-0432.CCR-17-1117. Epub 2017 Aug 1. PMID 28765323
- [Background] Osler M, Rozing MP, Christensen GT, Andersen PK, Jorgensen MB. Electroconvulsive therapy and risk of dementia in patients with affective disorders: a cohort study. Lancet Psychiatry. 2018 Apr;5(4):348-356. doi: 10.1016/S2215-0366(18)30056-7. Epub 2018 Mar 6. PMID 29523431
- [Background] Peterchev AV, Wagner TA, Miranda PC, Nitsche MA, Paulus W, Lisanby SH, Pascual-Leone A, Bikson M. Fundamentals of transcranial electric and magnetic stimulation dose: definition, selection, and reporting practices. Brain Stimul. 2012 Oct;5(4):435-53. doi: 10.1016/j.brs.2011.10.001. Epub 2011 Nov 1. PMID 22305345
- [Background] Phelps DL, Balog J, Gildea LF, Bodai Z, Savage A, El-Bahrawy MA, Speller AV, Rosini F, Kudo H, McKenzie JS, Brown R, Takats Z, Ghaem-Maghami S. The surgical intelligent knife distinguishes normal, borderline and malignant gynaecological tissues using rapid evaporative ionisation mass spectrometry (REIMS). Br J Cancer. 2018 May;118(10):1349-1358. doi: 10.1038/s41416-018-0048-3. Epub 2018 Apr 19. PMID 29670294
- [Background] Reid B, Zhao M. The Electrical Response to Injury: Molecular Mechanisms and Wound Healing. Adv Wound Care (New Rochelle). 2014 Feb 1;3(2):184-201. doi: 10.1089/wound.2013.0442. PMID 24761358
- [Background] Sawhney JP, Kothiwale VA, Bisne V, Durgaprasad R, Jadhav P, Chopda M, Vanajakshamma V, Meena R, Vijayaraghavan G, Chawla K, Allu J, Pieper KS, John Camm A, Kakkar AK; GARFIELD-AF Investigators. Risk profiles and one-year outcomes of patients with newly diagnosed atrial fibrillation in India: Insights from the GARFIELD-AF Registry. Indian Heart J. 2018 Nov-Dec;70(6):828-835. doi: 10.1016/j.ihj.2018.09.001. Epub 2018 Sep 12. PMID 30580852
- [Background] Strauch B, Herman C, Dabb R, Ignarro LJ, Pilla AA. Evidence-based use of pulsed electromagnetic field therapy in clinical plastic surgery. Aesthet Surg J. 2009 Mar-Apr;29(2):135-43. doi: 10.1016/j.asj.2009.02.001. PMID 19371845
- See also: Related Info — https://opendata.ncats.nih.gov/covid19/